CLINICAL TRIAL: NCT06811207
Title: Comparison of the Efficacies of Two Novel Dose Dual Therapies in the First-line Helicobacter Pylori Eradication
Acronym: Helicobacter
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 202200416A3; CMRPG8M1121 (Other Grant/Funding Number: Chang Gung Memorial Hospital)
Record Dates: First submitted 2024-11-19; First posted 2025-02-06 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-02

CONDITIONS: HELICOBACTER PYLORI INFECTIONS
Keywords: Helicobacter pylori; Potassium-competitive acid blocker; Proton pump inhibitors; High-dose dual therapy; Antibiotic susceptibility
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Esomeprazole; Amoxicillin

STUDY DESIGN:
Intervention Model Description: The investigators will recruit 300 adult participants with H. pylori infection from Kaohsiung Chang Gung Memorial Hospital. Using a computer-generated randomized sequence, we randomly allocated 150 patients to either 14-day high-dose dual therapy (vonoprazan 20 mg bid, and amoxicillin 750mg qid. for 14 days) or 150 participants (Esomeprezole 40 mg tid, and amoxicillin 750mg qid. for 14 days). Participants are asked to return in the second week to assess drug compliance and adverse events. Post-treatment H. pylori status is assessed by a 13C-urea breath test at week 8. Additionally, antibiotic susceptibility of H. pylori will be examined. Finally, the rates of eradication, adverse events, and compliance will be compared between two groups by chi-square test, and the host and bacterial factors influencing each efficacy of the regimen are assessed by multivariate analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 14-day PCAB-based high-dose dual therapy. (Active Comparator): vonoprazan 20 mg bid, and amoxicillin 750mg qid. for 14 days
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin
- 14-day PPI-Based High-Dose Dual Therapies (Experimental): Esomeprezole 40 mg tid, and amoxicillin 750mg qid. for 14 days
  Interventions: Drug: Esomeprazole 40mg; Drug: Amoxicillin

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan (20 mg bid, for 14 days)
  Arms: 14-day PCAB-based high-dose dual therapy.
Drug: Esomeprazole 40mg — Esomeprazole (40 mg tid, for 14 days)
  Arms: 14-day PPI-Based High-Dose Dual Therapies
Drug: Amoxicillin — Amoxicillin (750 mg qid, for 14 days)

SUMMARY:
Background:

The key factors for success are the maintenance of intragastric pH > 6 and the drug resistance to antibiotics. Proton pump inhibitor (PPI)-based high-dose dual therapy is a novel anti-Helicobacter pylori (H. pylori) treatment. According to the investigators' previous study, the Esomeprazole-based high-dose dual therapy can achieve a higher eradication rate than standard triple therapy. The main reason for the high eradication rate was the use of high-dose esomeprazole which maintained 24-hour high intra-gastric pH. Another important reason was that investigators used only one antibiotic (Amoxicillin) with very low antibiotic resistance rates (0-2%). As compared to quadruple concomitant therapy which uses 3 antibiotics (clarithromycin, amoxicillin, and metronidazole), concomitant therapy could induce drug resistance which could affect public health issues.

Vonoprazan is a new gastric acid suppression agent, classified as a potassium-competitive acid blocker (PCAB). Its acid inhibition efficacy is superior to that of PPI. It has been evidenced that 7-day vonoprazan-based triple therapy achieved a higher eradication rate than 7-day PPI-based triple therapy in the first-line treatment of H. pylori infection but vonoprazan-based high-dose dual therapy can achieve a higher eradication rate than PPI-based thigh-dose dual therapy remains unclear.

Aims: (1) To test whether the efficacies of 14-day PCAB-based high-dose dual therapy can achieve a higher eradication rate than 14-day PPI-based high-dose dual therapy in the first-line treatment of H. pylori infection, (2) to examine the impacts of antibiotic resistance of H. pylori on the eradication efficacies of these two high-dose dual anti- H. pylori treatments.

Methods: The investigators will recruit 300 adult participants with H. pylori infection from Kaohsiung Chang Gung Memorial Hospital. Using a computer-generated randomized sequence, the investigators randomly allocated 150 patients to either 14-day high-dose dual therapy (vonoprazan 20 mg bid, and amoxicillin 750mg qid. for 14 days) or 150 patients (Esomeprezole 40 mg tid, and amoxicillin 750mg qid. for 14 days). Participants are asked to return in the second week to assess drug compliance and adverse events. Post-treatment H. pylori status is assessed by a 13C-urea breath test at week 8. Additionally, antibiotic susceptibility of H. pylori will be examined. Finally, the rates of eradication, adverse events and compliance will be compared between two groups by chi-square test, and the host and bacterial factors influencing each efficacy of the regimen are assessed by multivariate analysis.

Expected results: The acid inhibition efficacy of PCAB is superior to that of PPI. The investigators expect the PCAB-based high-dose dual therapy can achieve a better H. pylori eradication rate the PPA-based high-dose dual therapy. Minor adverse effects can be expected in each group of participants.

ELIGIBILITY:
Inclusion Criteria:

1. At least 20 years of age, with endoscopically proven peptic ulcer diseases or gastritis are prospectively recruited for this pilot study

Exclusion Criteria:

1. Previous H. pylori-eradication therapy,
2. Ingestion of antibiotics, bismuth, or PPIs within the prior 4 weeks,
3. Patients with an allergic history to the medications used,
4. Patients with previous gastric surgery,
5. The coexistence of serious concomitant illness (for example, decompensated liver cirrhosis, uremia),
6. Pregnant women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants With Eradication of H. pylori Confirmed by Urea Breath Test (UBT) | 6 to 8 weeks after the completion of the 14-day treatment period.
  1. Description: This outcome will measure the percentage of participants in each treatment group (PCAB-based dual therapy and PPI-based dual therapy) who achieve H. pylori eradication.
  2. Definition of Eradication: Eradication is defined as a negative result on the Urea Breath Test (UBT).
  3. Calculation Method: The proportion of eradicated participants will be calculated as: (Number of participants with confirmed eradication by UBT) / (Total participants analyzed)×100%

SECONDARY OUTCOMES:
Association Between Antibiotic Resistance and H. pylori Eradication Rate | esistance testing at baseline, and eradication confirmation at 6 to 8 weeks post-treatment.
  1. Description: This outcome will evaluate whether pre-treatment antibiotic resistance (e.g., amoxicillin resistance) is associated with the eradication success rate of PCAB-based and PPI-based high-dose dual therapies.
  2. Statistical Analysis: The correlation between antibiotic resistance status (resistant vs. susceptible) and eradication outcome (eradicated vs. not eradicated) will be analyzed using appropriate logistic regression models or chi-square tests.

OTHER OUTCOMES:
Antibiotic Resistance Profile of H. pylori Prior to Treatment | Baseline (prior to treatment initiation).
  1. Description: This outcome will assess the pre-treatment antibiotic resistance of H. pylori strains collected from participants.
  2. Resistance Measurement: Resistance to amoxicillin and other relevant antibiotics will be determined through bacterial culture and susceptibility testing (e.g., MIC values in μg/mL or resistant/susceptible categories).

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Others, Taiwan

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data (IPD) from this study. The data include sensitive information that may compromise participant privacy, even if de-identified. Ethical considerations and privacy regulations prevent data sharing.

REFERENCES:
- [Background] Liu L, Shi H, Shi Y, Wang A, Guo N, Li F, Nahata MC. Vonoprazan-based therapies versus PPI-based therapies in patients with H. pylori infection: Systematic review and meta-analyses of randomized controlled trials. Helicobacter. 2024 May-Jun;29(3):e13094. doi: 10.1111/hel.13094. PMID 38790090
- [Background] Gotoda T, Kusano C, Suzuki S, Horii T, Ichijima R, Ikehara H. Clinical impact of vonoprazan-based dual therapy with amoxicillin for H. pylori infection in a treatment-naive cohort of junior high school students in Japan. J Gastroenterol. 2020 Oct;55(10):969-976. doi: 10.1007/s00535-020-01709-4. Epub 2020 Jul 14. PMID 32666199
- [Derived] Tai WC, Lu LS, Yang SC, Wang HM, Wu CK, Yao CC, Huang PY, Lee YC, Chuah SK, Liang CM. Comparative efficacy and safety of vonoprazan versus esomeprazole-based high-dose dual therapies for first-line Helicobacter pylori eradication: a randomized controlled trial. Therap Adv Gastroenterol. 2025 Sep 20;18:17562848251378066. doi: 10.1177/17562848251378066. eCollection 2025. PMID 40984972